CLINICAL TRIAL: NCT00755599
Title: The EASE Trial: Eisenhower's Alternative Speculum Examination
Brief Title: Eisenhower's Alternative Speculum Examination
Acronym: EASE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruiting issues
Sponsor: Eisenhower Army Medical Center (U.S. Federal Agency)
Collaborators: Pearl Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: DDEAMC 07-15
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Papanicolaou Smear
Keywords: Papanicolaou Smear; Vaginitis; Patient Satisfaction
MeSH Terms: conditions — Vaginitis; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomization into one of two arms
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- No Stirrups (Active Comparator): Vaginal speculum examinations done without stirrups. The woman's feet will be placed onto the exam table allowing maximal repositioning by the woman.
  Interventions: Procedure: no-stirrup vaginal examination
- Stirrups (Active Comparator): Speculum examination with feet in stirrups. The woman's feet will be placed into obstetric stirrups which fix the feet in place.
  Interventions: Procedure: Vaginal speculum examination done with stirrups.

INTERVENTIONS:
Procedure: no-stirrup vaginal examination — Vaginal speculum examination done with feet on table extender.
  Arms: No Stirrups
Procedure: Vaginal speculum examination done with stirrups. — Speculum examination done with feet in stirrups.
  Arms: Stirrups

SUMMARY:
This study will determine patient and provider preferences regarding vaginal speculum examinations done with and without stirrups.

Primary research hypothesis: Women undergoing speculum examination will experience at least 20% less physical discomfort, 20% less sense of vulnerability, and 20% less sense of loss of control when using a no-stirrup method of examination compared to traditional in-stirrup examinations.

Secondary research hypothesis: 25% or less of the providers taught this alternative method of speculum examination will find it to be unacceptable.

DETAILED DESCRIPTION:
Subjects will be consented for inclusion into the study at the time of their presentation for one of the eligible presenting complaints. Those that agree to be part of the study will then be randomized to either stirrup or no-stirrup examinations. This will be done by opening previously sealed envelops with a data collection sheet inside of it. The sheet will say "stirrups" or "no-stirrups" at the top. This choice will be made via a random number table prior to beginning the study. The patient will then undergo examination using the indicated procedure. See Appendix A.

All patients will undergo speculum examination with medium Graves speculum. Patients needing, or requesting, other size speculums will be removed from the study. The participating provider will fill out the top of the data collection sheets and the patient will be asked to fill out the bottom of the sheet after the provider leaves the room. The sheets will then be dropped off at the nurses' station or leave them in the examination room.

Multiple aspects of physical discomfort, sense of control and sense of vulnerability will be assessed using a continuous scale. Patients will be asked to place a mark on a continuous line between two extremes. The distance will then be measured in millimeters in order to convert it to a numeric value. The measurement will be done by an independent provider in a blinded manner.

Medical providers participating in the study will be consented for enrollment. They will be mailed consent forms and asked to sign them in front of a witness and mail the consent form back to the PI. They will be eligible as long as they believe they can enroll 25 patients over the course of approximately one year. Providers will be trained on how to perform a no-stirrup examination. The training will include standardized draping of patients as well as standardized positioning of patients in order to reduce the amount of variation introduced by the providers into these examinations. The training will include still images and an instructional video. The Principal Investigator will be available to anyone who has further questions regarding the technique. Participating providers will also be asked to perform at least 5 no-stirrup examinations on non-study subjects prior to beginning enrollment into the study to ensure familiarization with the technique. Providers will be recruited if they agree to attempt to enroll 25 or more patients to the study over the course of approximately one year. This will not be a difficult number to achieve for an active clinician.

Providers who had not been trained on the no-stirrup speculum examination prior to the beginning this study will be sent a questionnaire querying them about their experience with the method after all data is collected.

Protected Health Information will not be collect, so HIPAA forms will not be required.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older and able to consent for themselves. All women undergoing speculum examinations for the following list of reasons will be eligible for this study. No other reasons for speculum examinations will be eligible. Eligible reasons:
* Pap smears during well woman examinations
* Pap smears during routine early pregnancy visit
* vaginal discharge
* vaginal bleeding
* sexually transmitted disease check

Exclusion Criteria:

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
physical discomfort | Immediately post-procedure
  As measured by a visual analog scale immediately after the procedure.

SECONDARY OUTCOMES:
sense of loss of control | Immediately post-procedure
  As measured by a visual analog scale immediately after the procedure.
sense of vulnerability | Immediately post-procedure
  As measured by a visual analog scale immediately after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Dean A Seehusen, MD, MPH, Principal Investigator — Eisenhower Army Medical Center
Locations (1):
- Eisenhower Army Medical Center, Fort Gordon, Georgia, United States